CLINICAL TRIAL: NCT05612958
Title: Efficacy and Safety of a 'Graft/Prosthesis, Biomaterial (DKM410)' in the Treatment of Both Nasolabial Folds: Single Center, Prospective, Comparative, Randomized, Double Blinded (Subject, Evaluator), Matched Pairs Design, Non-inferiority, Pivotal Clinical Trial
Brief Title: Efficacy and Safety of a 'Graft/Prosthesis, Biomaterial (DKM410)' in the Treatment of Both Nasolabial Folds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dongkook Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DKM-410-MD-1
Record Dates: First submitted 2022-11-07; First posted 2022-11-10 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Nasolabial Folds

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DKM-410 (Experimental): Participants are injected with an appropriate amount(up to 2.0ml) depending on the degree of nasolabial folds at baseline
  Interventions: Device: DKM-410
- Juvederm ULTRA PLUS XC 1.0ml (Active Comparator): Participants are injected with an appropriate amount(up to 2.0ml) depending on the degree of nasolabial folds at baseline
  Interventions: Device: Juvederm ULTRA PLUS XC 1.0ml

INTERVENTIONS:
Device: DKM-410 — Injection up to 2.0ml
  Arms: DKM-410
Device: Juvederm ULTRA PLUS XC 1.0ml — Injection up to 2.0ml
  Arms: Juvederm ULTRA PLUS XC 1.0ml

SUMMARY:
The purpose of the study is to assess the efficacy and safety of a 'Graft/prosthesis, biomaterial (DKM410)' in the treatment of both nasolabial folds.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19 years and older
2. Wrinkle Severity Rating Scale (WSRS) 3 or 4
3. Visually symmetrical bilateral nasolabial folds
4. Agreed not to use any dermatological treatment and wrinkle-improving functional cosmetics.
5. Voluntarily decided to participate in the study and signed the informed consent form
6. Willing to follow the protocol

Exclusion Criteria:

1. History of undergoing a permanent or semi-permanent filler treatment on the face
2. Received soft tissue augmentation using HA filler or collagen for nasolabial folds within 18 months from screening.
3. Received any surgery or laser treatment, chemical filling, heart attack, or Botox injection within 24 weeks from the screening
4. History of allergic reactions to Hyaluronic Acid or Gram-positive bacteria protein
5. Hypersensitivity to Lidocaine or amide local anesthetic
6. Positive for the intradermal response test
7. History of severe or plurality of allergies
8. Having skin inflammation or infection in nasolabial folds
9. History of keloid formation, hyperpigmentation, or hypertrophic scars on the face.
10. History of streptococcal disease
11. Uncontrolled epilepsy
12. Porphyria
13. Having or being currently suffering from autoimmune diseases
14. History of immunodeficiency or immunosuppressive drugs
15. History of herpetic eruption
16. Having bleeding disorder or blood clotting disorder
17. Having anticoagulant drugs or components within 72 hours from the application of medical advice
18. Received antiplatelet drugs within 2 weeks from the application of medical advice
19. Having high dose vitamin E or nonsteroidal anti-inflammatory drugs (NSAIDs) and high dose vitamin C within one week from the application of medical advice
20. Received drugs that inhibit or decrease liver metabolism
21. Clinically significant abnormalities on electrocardiogram
22. Pregnant or breast-feeding or who planning to conceive
23. Clinically severe cardiovascular, digestive, respiratory, endocrine, central nervous system disorders or mental illness
24. Other investigational products or procedures within 3 months from screening
25. Not eligible due to other reasons at the investigator's discretion

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Change in WSRS(Wrinkle Severity Rating Scale) score by independent evaluators from Baseline to Week 24. | Baseline and Week 24
  Independent evaluators evaluate the WSRS score change at Week 24 compared to baseline.

SECONDARY OUTCOMES:
Change in Wrinkle Severity Rating Scale(WSRS) score by independent evaluators from Baseline to Weeks 8, 16 and 48. | Baseline and Weeks 8, 16 and 48.
  WSRS(Wrinkle Severity Rating Scale) grading scale from 1 to 5, with grade 1 as absent, grade 2 as mild, grade 3 as moderate, grade 4 as severe, grade 5 as extreme.
Success rate of treatment(N%) by independent evaluators from Baseline to Weeks 8, 16, 24 and 48. | Baseline and Weeks 8, 16, 24 and 48.
  The percentage of subjects whose WSRS score was lowered by 1 or more points.
Change in Wrinkle Severity Rating Scale(WSRS) score by investigator from Baseline to Weeks 8, 16, 24 and 48. | Baseline and Weeks 8, 16, 24 and 48.
  WSRS(Wrinkle Severity Rating Scale) grading scale from 1 to 5, with grade 1 as absent, grade 2 as mild, grade 3 as moderate, grade 4 as severe, grade 5 as extreme.
Success rate of treatment(N%) by investigator from Baseline to Weeks 8, 16, 24 and 48. | Baseline and Weeks 8, 16, 24 and 48.
  The percentage of subjects whose WSRS score was lowered by 1 or more points.
Global Aesthetic Improvement Scale (GAIS) from Baseline to Weeks 8, 16, 24 and 48. | Baseline and Weeks 8, 16, 24 and 48.
  Global Aesthetic Improvement Scale (GAIS) from -1 to 3, with grade -1 as worse, grade 0 as no change, grade 1 as improved, grade 2 as much improved, grade 3 as very much improved.
Visual Analog Scale (VAS) after the treatment. | Baseline
  Visual Analog Scale (VAS) from 0mm to 100mm, with 0mm as no pain, 100mm as maximum pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-Ang University Hospital, Seoul, South Korea